CLINICAL TRIAL: NCT04740489
Title: A Pilot Study Examining Participants Psychosocial Health, Physical Activity and Staff Experiences: Is Adapted Home-based Phase 3 Cardiac Rehabilitation Feasible and Beneficial?
Brief Title: The Impact of Covid-19 on Cardiac Rehabilitation Participants and Staff
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ant Shepherd (Other)
Collaborators: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Ant Shepherd, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Organization: University of Portsmouth (Other)
Other Study IDs: 005
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Phase 3 Cardiac rehabilitation — Phase 3 CR is a comprehensive outpatient programme, considered the core rehabilitation phase, in which participants receive structured exercise, health education, risk factor modification and psychological support. Upon discharge from clinically supervised phase 3 CR participants are generally signposted to long-term community-based exercise classes (phase 4). The current study will take place within a core phase 3 CR programme in the UK.

SUMMARY:
What are the experiences of staff and participants in phase 3 cardiac rehabilitation during the Covid-19 pandemic, and what impacts have adapted delivery had on participants' physical activity levels, mental health and well-being?

Cardiac rehabilitation (CR) is a vital service for individuals diagnosed and treated for cardiovascular disease (e.g., heart attack, angina, valve disease). The service helps to improve recovery rates through supporting patients with beneficial lifestyle changes (e.g., physical activity, healthy eating), and coping with emotional distress following a traumatic cardiac event. The environment in which CR is being delivered has changed in response to the Covid-19 pandemic, including remote working practices, and in some instances postponing of rehabilitation. Despite the public health rationale for such measures, it is essential to consider the impact of adapted services on patient's mental health and physical activity participation, and to consider staff experiences in using remote working regimes. The current study aims to recruit staff and patients from phase 3 cardiac rehabilitation across Hampshire Hospitals Foundation Trust to explore their experiences of adapted services through a mixed methods study design. Staff and patients will be interviewed over the phone to explore experiences and impacts of Covid-19 with their rich in-depth viewpoints and stories. In addition, during an 8 week period of rehabilitation, patients will be asked to report and record their physical activity levels with diaries and accelerometers (a wrist worn device measuring movement), record their resting blood pressure and heart rate, and complete questionnaires to assess changes in mental health. This study could help to understand the impact of the pandemic on cardiac patients recovery and on staff's experiences implementing programme changes to assist in preparing for the future of CR post COVID 19.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) causes 17.9 million deaths globally each year, an estimated 31% of all deaths worldwide. Individuals diagnosed with CVD (e.g., acute coronary syndrome) are typically referred to cardiac rehabilitation (CR) following acute treatment (e.g. percutaneous coronary intervention) to facilitate both physical and psychological recovery, as well as an absolute risk reduction in cardiovascular mortality.

The timescale of CR can be divided into 4 interlinked phases. Phase 1 is marked by admission to hospital and acute care (e.g., revascularisation). Phase 2 is considered as early rehabilitation following patient discharge, usually a period of 2-6 weeks home-based support (e.g., Heart Manual) depending on when a participant is considered fit enough to start a structured exercise programme. Phase 3 CR is a comprehensive outpatient programme, considered the core rehabilitation phase, in which participants receive structured exercise, health education, risk factor modification and psychological support. Upon discharge from clinically supervised phase 3 CR participants are generally signposted to long-term community based exercise classes (phase 4).

The current study will take place within a core phase 3 CR programme in the UK. According to the National Audit of CR, 75.4% of participants receive group-based supervised programmes, and only 8.8% of participants receive home-based services in the UK (BHF, 2019). Nevertheless, the environment in which CR is being delivered has dramatically changed in response to the COVID 19 pandemic. Staff have been redeployed to COVID units, limiting operative capabilities, and in some instances postponed rehabilitation. In the midst of this global crisis, The European Association of Preventive Cardiology recommended an increased patient turnover in CR, adoption of precautions during programmes (e.g., avoiding group exercises), shortening the programmes, and following participants with remote assessment. Despite the public health rationale for such measures, it is essential to consider the impact of adapted services on participant's psychosocial health and physical activity participation, and to consider staff experiences of adaptation 'on the fly' through remote working protocols.

An integral characteristic of group-based CR settings is a positive, supporting and inclusive climate that encourages participants to manage their emotions and illness perceptions to improve coping and recovery following a cardiac event . Currently, these interpersonal dynamics have dramatically altered with the shift to remote delivery of CR components (e.g., telephone, video, internet, and social media). Hence, some of the benefits of group and face to face rehabilitation have arguably been removed. In addition, participants are now having to cope with the added threat of catching COVID 19 and having to deal with some of the potentially distressing consequences of quarantine, such as post-traumatic stress symptoms, confusion and anger. Therefore, the CR work force needs to be resilient and innovative to support participants throughout the pandemic with home-based programmes and telemedicine.

Fortunately, there is an evidence base to suggest that home-based programmes, such as the "Heart Manual", are as effective as centre-based CR in improving clinical and health-related quality of life outcomes. Indeed, novel interventions, such as telehealth weight management, Rehabilitation EnAblement in Chronic Heart Failure (REACH-HF), and cardiac telerehabilitation interventions, such as REMOTE-CR, are effective alternatives to the 'gold standard' centre-based provision. However, these findings are typically based upon randomised controlled trials (RCT) and are rarely investigated within real-world clinical settings where the research to practice gap needs to be negotiated. Scaling up RCT's and implementing novel remote programmes into CR promptly and effectively during the current pandemic could be a challenging process impacted by attitudes towards change, resources available, expertise, time, and competing priorities. Hence, it is important to assess and understand the real-world patient outcomes (e.g., physical activity participation, psychosocial and physical health) and the complexity of employing adapted CR services during the Covid-19 pandemic, including the barriers and facilitators to such implementation.

The purpose of this pilot study is to obtain quantitative and qualitative data to:

1. Assess the impact of adapted CR modalities in the UK on participants' physiological health, psychosocial health and physical activity behaviour
2. Explore CR staff's experiences of adapted delivery
3. Determine the feasibility of an adapted home-based CR programme for routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Staff and participants participating in Phase 3 CR
* Able to give informed consent
* Willing and able to undertake the interview, diary, questionnaire and accelerometer processes

Exclusion Criteria:

* Aged <18 years
* Not participating in Phase 3 CR
* Any individuals who are unable to represent their own interests or are particularly susceptible to coercion (vulnerable individuals), and are therefore unable to give informed consent
* If individuals have difficulties in adequately understanding written or verbal information in English, as the study doesn't have funding for a translator or interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Service user participants are individuals treated for acute coronary syndromes (e.g., NSTEMI, STEMI), heart failure, valve disease, and ICD's.
  Staff participants will be recruited from members of a multidisciplinary team including; CR professionals including CR specialist nurses, physiotherapists and exercise practitioners.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Psychosocial health and wellbeing | During qualitative interviews (post week 5).
  Semi structured interviews

SECONDARY OUTCOMES:
Acceptability to Participants | During qualitative interviews after the intervention has ended (post week 5).
  Qualitative interviews
Feasible to Participants | During qualitative interviews after the intervention has ended (post week 5).
  Qualitative interviews
Physical activity | Week 1, 4 and 8 of rehabilitation
  Accelerometer
Loneliness | Week 1, 4 and 8 of rehabilitation
  University of California, Los Angeles (UCLA) loneliness scale version 3 (minimum score 20 maximum of 80). Higher score signifies more loneliness
Heart rate | Week 1, 4 and 8 of rehabilitation
  Beats per minute
Blood pressure | Week 1, 4 and 8 of rehabilitation
  mmHg
Disease management | Week 1, 4 and 8 of rehabilitation
  Patient activation measure (Questionnaire)
Disease management | Week 1, 4 and 8 of rehabilitation
  The Cardiac Self-Efficacy (CSE) Scale. (minimum score 0 maximum of 52). Higher score indicates higher cardiac self-efficacy

IPD SHARING:
Plan to Share IPD: Undecided
Physical data will be made available. Interview transcripts will not as participants could be identified.